CLINICAL TRIAL: NCT03726112
Title: A Randomized, Double Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of SpotOn Specs for the Treatment of Chronic Dizziness & Imbalance
Brief Title: Spoton Trial Evaluating the Efficacy on BAlance Disorder sYmptoms (STEADY)
Acronym: STEADY
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Under internal considerations
Sponsor: SpotOn Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SpotOn_02
Record Dates: First submitted 2018-10-15; First posted 2018-10-31 (Actual); Last update posted 2019-05-08 (Actual); Status verified 2019-05

CONDITIONS: Balance Disorders

STUDY DESIGN:
Intervention Model Description: A Randomized, Double Blind, Placebo-Controlled Study followed by an open label phase
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SpotOn Specs (Active Comparator): Eyeglasses with Neuro-Balance Active (NBA) Spots
  Interventions: Device: SpotOn Specs
- Sham Specs (Sham Comparator): Eyeglasses with spots placed in peripheral zones previously identified as neutral
  Interventions: Device: Sham Specs

INTERVENTIONS:
Device: SpotOn Specs — SpotOn Balance glasses consists of unique visual stimuli (SpotOn's Neuro Balance Active Spots) applied to specific zones in the peripheral visual field
  Arms: SpotOn Specs
Device: Sham Specs — Sham device
  Arms: Sham Specs

SUMMARY:
A Randomized, Double Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of SpotOn specs for the Treatment of Chronic Dizziness & Imbalance.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18≤ years ≤70
* DHI score of at least 36 (moderate to severe handicap)
* One or more symptoms of unsteadiness, dizziness or vertigo are present on most days. Symptoms could vary in intensity however lasts for 3 months or more
* Ability to perform all tests (including computerized test) and interviews
* At least three months after the last Vestibular Balanced Rehabilitation Therapy - (if applicable)
* Gave informed consent for participation in the study

Exclusion Criteria:

* Dizziness disease with fluctuating symptoms
* Any active or non-controlled disease that might cause dizziness and imbalance, unless well controlled for at least 3 months
* Moderate-Severe Depression or Anxiety
* Known related eye disease
* Pregnant women
* Currently taken part in a clinical trial or within 30 days prior to screening
* Concomitant use of any medications that might affect the balance system

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Dizziness Handicap Inventory (DHI) | baseline, 8 weeks
  The Dizziness Handicap Inventory (DHI) is a 25-item self-assessment scale. A "yes" response to an item is awarded 4 points, a "sometimes" 2 points, and a "no", 0 points. Possible scores on the DHI range from 0 (suggesting no handicap) to 100, indicating significant perceived handicap

SECONDARY OUTCOMES:
Clinical Global Impression of Improvement | 8 weeks
  The Clinical Global Impression scale is a clinician-rated scale used to rate patients' improvement from baseline, based on the subject's baseline status- Improvement is rated on a scale of 1-7, with 1 being "very much improved" and 7 being "very much worse"
Change from baseline in the Clinical Global Impression of Severity | baseline, 8 weeks
  A clinician-rated scale used to rate patients' severity of symptoms. Severity is rated on a scale of 1-7 with one being "normal, not at all ill," and 7 being "among the most extremely ill patients."
Change from baseline in Postural sway | baseline, 8 weeks
  Postural control will be measure during stance and gait
Change from baseline in the Visual Vertigo Analog Scale (VVAS) | baseline, 8 weeks
  A visual analogue scale subjects are asked to evaluate their subjective feeling of dizziness in the last week on a scale from 0 (no dizziness at all) to 10 (very severe dizziness)
Change from baseline in the Beck Anxiety Inventory | baseline, 8 weeks
  A self-report inventory for measuring the severity of an individual's anxiety. The BAI contains 21 questions, each answer being scored on a scale value of 0 (not at all) to 3 (severely). Higher total scores indicate more severe anxiety symptoms.
Change from baseline in the Vertigo Symptom Scale-Short Form (VSS-SF) | baseline, 8 weeks
  The VSS assesses symptoms of balance system dysfunction (for example, dizziness, vertigo, postural instability, and falling) and symptoms of somatic anxiety and autonomic arousal (diverse pains and somatic sensations, sweating, pounding heart, breathing difficulties, and fainting). A measure of symptom severity is obtained by summing the item scores. The total scale score ranges 0-60, higher scores indicating more severe problems.
Incident rate of falls | 8 weeks
  Reported falls during the study

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Shlamkovitz, MD, Principal Investigator — Assaf Harofeh Medical Center, Rishon LeZion, ENT Department
Locations (1):
- Assaf Harofeh Medical Center, Rishon LeZion, ENT Department, Rishon LeZiyyon, Israel